CLINICAL TRIAL: NCT02100917
Title: Bioequivalence Study Evaluating the Pharmacokinetics of DMB-3111 and Trastuzumab in Healthy Japanese Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Collaborators: Dong-A Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DMB-3111-2; JapicCTI-142486 (Registry Identifier: Japan Primary Registries Network)
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Volunteer
Keywords: Bioequivalence; Biosimilarity; Similarity; Pharmacokinetics; Phase I; Trastuzumab; Healthy Male Volunteers; Single-dose; HER-2; Oncology
MeSH Terms: conditions — Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMB-3111 (Experimental): 6 mg/kg is once given in intravenous drip infusion taking 90 min
  Interventions: Drug: DMB-3111
- trastuzumab (Active Comparator): 6 mg/kg is once given in intravenous drip infusion taking 90 min
  Interventions: Drug: trastuzumab

INTERVENTIONS:
Drug: DMB-3111
  Arms: DMB-3111
Drug: trastuzumab
  Arms: trastuzumab

SUMMARY:
This study is a randomized Trastuzumab-controlled double-blind parallel-group study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese male adults
2. Body Mass Index (BMI) between 17.6 and 26.4 kg/m² at the time of screening BMI = Body Weight (kg)/[Height (m)]²
3. The individual who freely consents to participate after receiving a detailed explanation of the clinical study and completely understanding thereof, and who has capacity to follow precautions and provide written consent.

Exclusion Criteria:

1. History of hypersensitivity to components of Trastuzumab or diphenhydramine or any other drug
2. Use of any ethical drug within 2 weeks before investigational product administration or any over-the-counter drug within 1 week before investigational product administration that would affect study participation in the opinion of the investigator or subinvestigators (except for diphenhydramine, which will be used concomitantly in the present clinical trial and any drug applied locally and having no systemic actions)
3. History of allergic symptoms such as bronchial asthma and urticaria that would affect study participation in the opinion of the investigator or subinvestigators
4. History of cardiac disorders, hypertension, coronary artery disease (e.g., myocardial infarction, angina), and/or vascular disorder; ongoing palpitations, shortness of breath, and/or tachycardia

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time (AUC) | Day1-71
Maximum observed serum concentration (Cmax) | Day1-71

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) from 0 to time of the last measurable concentration | Day1-71
Area under the concentration-time curve (AUC) from 0 to infinity | Day1-71
Time to reach the peak concentration (tmax) | Day1-71
Mean residence time (MRT) from 0 to final sampling time point | Day1-71
Mean residence time (MRT) from 0 to infinity | Day1-71
elimination rate constant (kel) | Day1-71
Elimination half life (t1/2) | Day1-71
Clearance (CL) | Day1-71
Incidence of adverse events | Day1-71

OTHER OUTCOMES:
Incidence of anti-trastuzumab antibodies (ADAs) | Day1-71

CONTACTS AND LOCATIONS:
Locations (1):
- Fukuoka, Fukuoka, Japan

REFERENCES:
- [Derived] Morita J, Tanaka M, Nomoto M, Matsuki S, Tsuru T, Matsuguma K, Shiramoto M. Pharmacokinetic Bioequivalence, Safety, and Immunogenicity of DMB-3111, a Trastuzumab Biosimilar, and Trastuzumab in Healthy Japanese Adult Males: Results of a Randomized Trial. BioDrugs. 2016 Feb;30(1):17-25. doi: 10.1007/s40259-015-0153-2. PMID 26691837